CLINICAL TRIAL: NCT00265304
Title: A Double-Blind, Long-Term Evaluation of the Safety of IDEA-033 in Comparison to Oral Naproxen for the Treatment of the Signs and Symptoms of Osteoarthritis of the Knee
Brief Title: A Long-Term Safety Study of IDEA-033 in Comparison to Oral Naproxen for the Treatment of Osteoarthritis of the Knee
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: IDEA AG (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CL-033-III-05; NCT00371358 (obsolete NCT alias)
Record Dates: First submitted 2005-12-13; First posted 2005-12-14 (Estimated); Last update posted 2009-03-20 (Estimated); Status verified 2009-03

CONDITIONS: Osteoarthritis, Knee
Keywords: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Ketoprofen

INTERVENTIONS:
Drug: Ketoprofen

SUMMARY:
The purpose of this study is to evaluate the long-term safety of IDEA-033 (an anti-inflammatory pain-relieving drug applied to the skin) in comparison to naproxen (an anti-inflammatory pain-relieving drug taken by mouth) for the treatment of osteoarthritis of both knees.

DETAILED DESCRIPTION:
This is a double-blind, active-controlled study of the safety of IDEA-033 in comparison to oral naproxen for the treatment of the signs and symptoms of osteoarthritis of the knee in patients who have completed Study 17-007 or who have discontinued Study 17-007 due to lack of efficacy. If a sufficient number of patients do not enroll from Study 17-007, patients with osteoarthritis of both knees who were not enrolled in Study 17-007 may be enrolled in this study. Patients treated with IDEA-033 in Study 17-007 will receive 100 mg per knee of ketoprofen gel twice daily and one placebo capsule twice daily for 52 weeks. Patients treated with oral naproxen or placebo in Study 17-007 will receive a 500 mg naproxen over-encapsulated tablet twice daily and placebo topical gel twice daily for 52 weeks. Patients who did not participate in Study 17-007 will be randomized to receive one of these two treatments. The primary outcomes of the study include the incidence and severity of adverse events, dermal-irritation scores, and changes in routine clinical laboratory tests and vital signs obtained at each visit.

Patients assigned to IDEA-033 in Study 17-007 will topically apply 100 mg per knee of ketoprofen gel twice daily and take one oral placebo capsule twice daily for 52 weeks. Patients assigned to oral naproxen or placebo in Study 17-007 will take one 500 mg naproxen over-encapsulated tablet orally twice daily and apply placebo topical gel twice daily for 52 weeks. Patients who did not participate in Study 17-007 will be randomized to receive one of these two treatments.

ELIGIBILITY:
Inclusion Criteria:

* Patients who completed Study 17-007 or discontinued from Study 17-007 due to lack of efficacy
* Patients who did not complete or discontinue from Study 17-007 must have osteoarthritis of both knees for a minimum of six months
* Have moderate pain in the most involved knee when not taking non-steroidal anti-inflammatory drugs (NSAIDs)
* Must have used an oral NSAID on at least three days per week for the last three months, or 25 of the 30 days before screening
* Demonstrate x-ray evidence of osteoarthritis in the most involved knee during the last six months

Exclusion Criteria:

* Any patient currently receiving physical therapy to either knee or having a history of allergy, hypersensitivity or contraindication to ketoprofen, naproxen, or acetaminophen, an NSAID idiosyncrasy, or any other medical condition that would compromise the ability of the subject to complete the required assessments and visits
* For patients who did not participate in Study 17-007: having Grade 1 or Grade 4 severity of the most involved knee based on x-ray criteria
* Received intra-articular injections or arthroscopy of the most involved knee during three months before screening visit
* Have a large bulging effusion, or have inflammation of the most involved knee that could be related to gout, pseudogout-induced synovitis, or infection
* Have a history of partial or total knee replacement in either knee, or have a history of gout, pseudo-gout induced synovitis, or infection of the more severe knee

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550
Dates: Start 2005-07; Primary Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Adverse events; Dermal-irritation scores; Changes in routine clinical laboratory tests and vital signs obtained at each visit.

SECONDARY OUTCOMES:
Change from baseline (Week 12 for patients who completed 17-007, baseline for those who did not) and mean value per visit for WOMAC pain, stiffness, and physical function scores; Subject Global Assessment of Response to Therapy.

CONTACTS AND LOCATIONS:
Overall Officials: IDEA AG Clinical Trial, Study Director — IDEA AG
Locations (82):
- United States (82):
  - Capstone Clinical Trials Inc, Birmingham, Alabama
  - Montgomery, Alabama
  - Northport, Alabama
  - Mesa, Arizona
  - Phoenix, Arizona
  - Tempe, Arizona
  - Anaheim, California
  - Encinitas, California
  - Fair Oaks, California
  - Garden Grove, California
  - Irvine, California
  - Paramount, California
  - Rancho Mirage, California
  - San Diego, California
  - Spring Valley, California
  - Vista, California
  - Northglenn, Colorado
  - Danbury, Connecticut
  - Clearwater, Florida
  - Coral Gables, Florida
  - Radiant Research-daytona, Daytona Beach, Florida
  - DeLand, Florida
  - Fort Myers, Florida
  - Gainesville, Florida
  - The Community Research of South Florida, Hialeah, Florida
  - Ocala, Florida
  - Ocoee, Florida
  - Palm Harbor, Florida
  - Pembroke Pines, Florida
  - Port Orange, Florida
  - Tampa, Florida
  - West Palm Beach, Florida
  - International Research Center, Atlanta, Georgia
  - Atlanta, Georgia
  - Evansville, Indiana
  - Arkansas City, Kansas
  - Newton, Kansas
  - Wichita, Kansas
  - Louisville, Kentucky
  - Milford, Massachusetts
  - East Lansing, Michigan
  - Kalamazoo, Michigan
  - Lansing, Michigan
  - Flowood, Mississippi
  - Jackson, Mississippi
  - Bozeman, Montana
  - Las Vegas, Nevada
  - Berlin, New Jersey
  - Dover, New Jersey
  - Binghamton, New York
  - Manilus, New York
  - Rochester, New York
  - Durham, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Community Research Managment Associates, Cincinnati, Ohio
  - Columbus, Ohio
  - Franklin, Ohio
  - Perrysburg, Ohio
  - Gilbert Medical Research, Bethany, Oklahoma
  - Beaver, Pennsylvania
  - Bensalem, Pennsylvania
  - Duncansville, Pennsylvania
  - Harleysville, Pennsylvania
  - Levittown, Pennsylvania
  - Penndel, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Warwick, Rhode Island
  - Anderson, South Carolina
  - Charleston, South Carolina
  - Columbia, South Carolina
  - Greer, South Carolina
  - Memphis, Tennessee
  - Austin, Texas
  - Dallas, Texas
  - Houston, Texas
  - Lake Jackson, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Spokane, Washington
  - Glendale, Wisconsin